CLINICAL TRIAL: NCT00866723
Title: Phase II Study of Single-Agent Avastin in Patients With Epithelial Ovarian, Primary Peritoneal Serous, Papillary Serous Endometrial or Fallopian Tube Cancer Who Have Recurred After Prior Therapy With Maintenance Avastin
Brief Title: Avastin in Patients With Epithelial Ovarian, Primary Peritoneal Serous or Fallopian Tube Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment has been terminated prematurely because of poor enrollment.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Panagiotis Konstantinopoulos, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-323
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Serous Cancer; Fallopian Tube Cancer
Keywords: Avastin; bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab (Experimental): Bevacizumab was administered at 15 mg/kg intravenously every 3 weeks. Treatment continued until disease progression or unacceptable toxicity.
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of this study is to evaluate how the participant's disease (ovarian, primary peritoneal serous, fallopian tube, or papillary serous endometrial cancer) responds to additional treatment with Avastin (bevacizumab). Participants have already received Avastin as part of maintenance therapy for their cancer. Maintenance therapy is a medical therapy that is given to people to prevent a relapse. However, cancer may return after maintenance therapy. This research study hopes to determine whether additional treatment with Avastin will be effective in treating the participant's cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

To determine the activity of bevacizumab in patients with epithelial ovarian, primary peritoneal serous, papillary serous endometrial or fallopian tube cancer who relapse after achieving an initial complete response to first-line therapy that included at least 6 month bevacizumab maintenance as defined by: 1) clinical response rate OR 2) clinical benefit response

Secondary:

* To assess duration of progression free survival (PFS)
* To assess the safety
* To correlate response with the Avastin-free interval

STATISTICAL DESIGN:

This study used a two-stage design to evaluate efficacy of bevacizumab based on a patient achieving either clinical response or clinical benefit response. The null and alternative response rates were 10% and 30%. If two or more patients enrolled in the stage one cohort (n=10 patients) achieved response than accrual would proceed to stage two (n=19 patients). If response was achieved by at least 6 patients in the final set of 29 evaluable patients then bevacizumab would be deemed worthy for further study. This design had 80% power given one-sided 0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed epithelial ovarian cancer, primary peritoneal serous cancer, papillary serous endometrial cancer, or fallopian tube cancer
* Must have responded and remained clinically stable (as defined by normal clinical examination, normal serum CA125 level and normal CT scan) after first-line platinum-based regimen followed by bevacizumab maintenance therapy
* Must have developed relapsed disease at least 3 months after completion of bevacizumab maintenance therapy as defined by a) development of new, measurable lesions by RECIST criteria, but no lesion with maximum diameter greater than 3 centimeters OR b) newly elevated CA125 level at least 2 x ULN on 2 separate occasions, obtained at least 1 day but not more than 3 months apart
* ECOG Performance Status 0-2
* No prior cytotoxic chemotherapy or biologic therapy for disease recurrence allowed
* Prior hormonal-based therapy for ovarian, primary peritoneal serous or fallopian tube cancer is allowed
* Toxic side effects related to prior chemotherapy or hormonal therapy must have resolved to grade one or less or to baseline before initiation of bevacizumab
* 18 years of age or older
* Life expectancy of 6 months or greater
* Normal organ and marrow function as outlined in the protocol

Exclusion Criteria:

* Prior cytotoxic chemotherapy or biologic therapy for disease recurrence
* Known CNS disease, except for treated brain metastasis
* Pregnancy or breast feeding
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0, or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular device, within 7 days prior to enrollment
* History of abdominal fistula, GI perforation, intra-abdominal abscess, or CT evidence of bowel obstruction or bowel wall thickening
* Symptoms of intestinal obstruction, or requirement of parenteral hydration and/or nutrition
* History of active malignancy during the last 3 years, except non-melanomatous skin cancer or in situ breast or cervical cancer
* Evidence of preexisting uncontrolled hypertension. If patient has hypertension, it must be medically controlled (< 150/90) prior to starting bevacizumab
* Proteinuria at screening
* Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent
* Therapeutic anticoagulation is not by itself and exclusion criterion. However, for certain high risk patients on therapeutic anticoagulation, eligibility will be determined after discussion with the overall PI
* Any active bleeding
* Serious, non-healing wound, ulcer, or bone fracture
* Prior history of hypertensive crisis or hypertensive encephalopathy
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to day 1
* Significant vascular disease within 6 months prior to day 1
* History of hemoptysis within 1 month prior to day 1
* Presence of measurable lesion(s) by RECIST criteria with maximum diameter greater than 3 centimeters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Result] Konstantinopoulos PA, Berlin ST, Campos SM, Matulonis UA, Cannistra SA. Bevacizumab rechallenge after first line maintenance bevacizumab. Gynecol Oncol. 2012 May;125(2):510-1. doi: 10.1016/j.ygyno.2012.02.013. Epub 2012 Feb 21. No abstract available. PMID 22366591

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab
Started | 5
Completed | 0
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 55 [38 to 68]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: For measurable disease (MD) patients, clinical response on treatment was based on RECIST 1.0 criteria with overall response defined as achieving partial response (PR) or complete response (CR). Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. For non-MD patients, clinical response based on modified Gynecologic Cancer Intergroup (GCIG) criteria was defined as at least a 50% decrease in CA-125 levels.
Time Frame: Disease was evaluated at baseline and every 3 cycles on treatment. Treatment continued until disease progression or unacceptable toxicity. Patients underwent radiologic assessment (CT or MRI scans) and CA-125 levels were measured.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
proportion of participants | 0.20 [0.01 to 0.66]

2. Primary Outcome: Clinical Benefit Response Rate
Description: Clinical benefit response was defined as absence of disease progression at 18 weeks (ie after 6 cycles). Disease progression (PD) could occur per RECIST 1.0 or based on CA-125 levels. Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Disease progression based on CA-125 level was doubling of the CA-125 level from baseline. For patients with normal baseline CA-125 (who by definition had MD) the criterion for progression based on CA-125 doubling was doubling of CA-125 from the upper limit of normal (i.e. more than 70).
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of particpants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
proportion of particpants | 0.80 [0.34 to 0.99]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. There were no SAEs experinced by patients on this study per the above definition.
  Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=5)
Hypertension (Vascular disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1
Chelitis (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No